CLINICAL TRIAL: NCT03088657
Title: Mood Disorder Cohort Research Consortium (MDCRC) in Korea
Brief Title: Design and Methods of the Mood Disorder Cohort Research Consortium (MDCRC) Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government); Seoul National University Hospital (Other); Severance Hospital (Other); Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other); Gyeongsang National University Hospital (Other); Pusan National University Hospital (Other); Chonnam National University Hospital (Other); National Center for Mental Health, Korea (Unknown)
Responsible Party: Principal Investigator, Heon-Jeong Lee, MD, PhD, Professor, Korea University Anam Hospital
Other Study IDs: MDCRC
Record Dates: First submitted 2017-03-03; First posted 2017-03-23 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Mood Disorders; Bipolar Disorder; Major Depressive Disorder
Keywords: Cohort study; early-onset mood disorders
MeSH Terms: conditions — Mood Disorders; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — blood 10cc
Oversight: Data Monitoring Committee: No

SUMMARY:
The Mood Disorder Cohort Research Consortium (MDCRC) study is designed as a naturalistic observational prospective cohort study for early-onset mood disorders (major depressive disorders, bipolar disorders type 1 and 2) in South Korea.

DETAILED DESCRIPTION:
The Mood Disorder Cohort Research Consortium (MDCRC) study is designed as a naturalistic observational prospective cohort study for early-onset mood disorders (major depressive disorders, bipolar disorders type 1 and 2) in South Korea. The study subjects consist of two populations: 1) patients with mood disorders under 25 years old and 2) patients with mood disorders within 2 years of treatment under 35 years old. After successful screening, the subjects are evaluated using baseline assessments and serial follow-up assessments at 3-month intervals. Between the follow-up assessments, subjects are dictated to check their own daily mood status before bedtime using the eMood chart application or a paper mood diary. In addition, wearable activity tracker(Fitbit charge series) is applied for data collection such as activity, sleep, and heart rate during every moments. At the regular visits every 3 months, inter-visit assessments are evaluated based on daily mood charts and interviews with patients. In addition to the daily mood chart, sleep quality, inter-visit major and minor mood episodes, stressful life events, and medical usage pattern with medical expenses are also assessed. Genomic DNA from blood is obtained for genomic analyses. From the MDCRC study, the clinical course, prognosis, and related factors of early-onset mood disorders can be clarified. The MDCRC is also able to facilitate translational research for mood disorders and provide a resource for the convergence study of mood disorders.

ELIGIBILITY:
Inclusion Criteria:

1. under 25 years old with mood disorder
2. under 35 years old with mood disorder within 2 years of treatment

Exclusion Criteria:

1. patients with intellectual disability
2. patients with organic brain injury
3. patients have difficulty reading and understanding the Korean language

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: mood disorder patients who fulfill the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) for major depressive disorder, bipolar I disorder, or bipolar II disorder
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-09; Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
illness severity and change in patients by using Clinical Global Impression-Bipolar score | 3months

SECONDARY OUTCOMES:
Scores of depressive symptoms as assessed by MADRS | 3months
  MADRS : Montgomery-Åsberg Depression Rating Scale
Scores of manic symptoms as assessed by YMRS | 3months
  YMRS : Young Mania Rating Scale
Daily mood chart | 3 months
  subjects are dictated to check their own daily mood status before bedtime using the eMood chart application or a paper mood diary. Patients are provided a daily mood chart that asks for mood state (-3 to +3), energy level (-3 to +3), anxiety (0-3), irritability (0-3).
Sleep | 3months
  Daily data from wearable device by using Fitbit charge series.
Activity | 3months
  Daily data from wearable device by using Fitbit charge series.
Heart rate | 3months
  Daily data from wearable device by using Fitbit charge series.
average monthly cost of treatment for psychiatric, medical, dental, and oriental medicinal management | 3months

CONTACTS AND LOCATIONS:
Overall Officials: Heon-Jeong Lee, MD, PhD, Principal Investigator — 'Korea University Anam Hospital' in Seoul, Korea
Locations (1):
- Heon-Jeong Lee, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho CH, Ahn YM, Kim SJ, Ha TH, Jeon HJ, Cha B, Moon E, Park DY, Baek JH, Kang HJ, Ryu V, An H, Lee HJ. Design and Methods of the Mood Disorder Cohort Research Consortium (MDCRC) Study. Psychiatry Investig. 2017 Jan;14(1):100-106. doi: 10.4306/pi.2017.14.1.100. Epub 2016 Dec 29. PMID 28096882
- [Result] Chang SM, Hong JP, Cho MJ. Economic burden of depression in South Korea. Soc Psychiatry Psychiatr Epidemiol. 2012 May;47(5):683-9. doi: 10.1007/s00127-011-0382-8. Epub 2011 Apr 28. PMID 21526429
- [Result] Murphy JA, Byrne GJ. Prevalence and correlates of the proposed DSM-5 diagnosis of Chronic Depressive Disorder. J Affect Disord. 2012 Jul;139(2):172-80. doi: 10.1016/j.jad.2012.01.033. Epub 2012 Mar 3. PMID 22381955
- [Result] Hunter AM, Leuchter AF, Morgan ML, Cook IA. Changes in brain function (quantitative EEG cordance) during placebo lead-in and treatment outcomes in clinical trials for major depression. Am J Psychiatry. 2006 Aug;163(8):1426-32. doi: 10.1176/ajp.2006.163.8.1426. PMID 16877657
- [Result] Tenke CE, Kayser J, Manna CG, Fekri S, Kroppmann CJ, Schaller JD, Alschuler DM, Stewart JW, McGrath PJ, Bruder GE. Current source density measures of electroencephalographic alpha predict antidepressant treatment response. Biol Psychiatry. 2011 Aug 15;70(4):388-94. doi: 10.1016/j.biopsych.2011.02.016. Epub 2011 Apr 20. PMID 21507383
- [Result] Iosifescu DV, Greenwald S, Devlin P, Perlis RH, Denninger JW, Alpert JE, Fava M. Pretreatment frontal EEG and changes in suicidal ideation during SSRI treatment in major depressive disorder. Acta Psychiatr Scand. 2008 Apr;117(4):271-6. doi: 10.1111/j.1600-0447.2008.01156.x. Epub 2008 Feb 26. PMID 18307587
- [Result] Chang JS, Yoo CS, Yi SH, Her JY, Choi HM, Ha TH, Park T, Ha K. An integrative assessment of the psychophysiologic alterations in young women with recurrent major depressive disorder. Psychosom Med. 2012 Jun;74(5):495-500. doi: 10.1097/PSY.0b013e31824d0da0. Epub 2012 Mar 9. PMID 22408133
- [Result] Suto T, Fukuda M, Ito M, Uehara T, Mikuni M. Multichannel near-infrared spectroscopy in depression and schizophrenia: cognitive brain activation study. Biol Psychiatry. 2004 Mar 1;55(5):501-11. doi: 10.1016/j.biopsych.2003.09.008. PMID 15023578
- [Result] Kromer SA, Kessler MS, Milfay D, Birg IN, Bunck M, Czibere L, Panhuysen M, Putz B, Deussing JM, Holsboer F, Landgraf R, Turck CW. Identification of glyoxalase-I as a protein marker in a mouse model of extremes in trait anxiety. J Neurosci. 2005 Apr 27;25(17):4375-84. doi: 10.1523/JNEUROSCI.0115-05.2005. PMID 15858064
- [Result] Paige LA, Mitchell MW, Krishnan KR, Kaddurah-Daouk R, Steffens DC. A preliminary metabolomic analysis of older adults with and without depression. Int J Geriatr Psychiatry. 2007 May;22(5):418-23. doi: 10.1002/gps.1690. PMID 17048218
- [Result] Yang Z, Ma X, Wang Y, Wang J, Xiang B, Wu J, Deng W, Li M, Wang Q, Li T. Association of APC and REEP5 gene polymorphisms with major depression disorder and treatment response to antidepressants in a Han Chinese population. Gen Hosp Psychiatry. 2012 Sep-Oct;34(5):571-7. doi: 10.1016/j.genhosppsych.2012.05.015. Epub 2012 Jul 12. PMID 22795047
- [Result] Kocabas NA. Catechol-O-methyltransferase (COMT) pharmacogenetics in the treatment response phenotypes of major depressive disorder (MDD). CNS Neurol Disord Drug Targets. 2012 May;11(3):264-72. doi: 10.2174/187152712800672445. PMID 22483292
- [Result] Dreimuller N, Tadic A, Dragicevic A, Boland K, Bondy B, Lieb K, Laux G, Maier W, Muller MJ, Rao ML, Rietschel M, Roschke J, Zill P, Hiemke C. The serotonin transporter promoter polymorphism (5-HTTLPR) affects the relation between antidepressant serum concentrations and effectiveness in major depression. Pharmacopsychiatry. 2012 May;45(3):108-13. doi: 10.1055/s-0031-1291347. Epub 2011 Nov 15. PMID 22086748
- [Derived] Lim D, Jeong J, Song YM, Cho CH, Yeom JW, Lee T, Lee JB, Lee HJ, Kim JK. Accurately predicting mood episodes in mood disorder patients using wearable sleep and circadian rhythm features. NPJ Digit Med. 2024 Nov 18;7(1):324. doi: 10.1038/s41746-024-01333-z. PMID 39557997
- [Derived] Cho CH, Lee T, Lee JB, Seo JY, Jee HJ, Son S, An H, Kim L, Lee HJ. Effectiveness of a Smartphone App With a Wearable Activity Tracker in Preventing the Recurrence of Mood Disorders: Prospective Case-Control Study. JMIR Ment Health. 2020 Aug 5;7(8):e21283. doi: 10.2196/21283. PMID 32755884